CLINICAL TRIAL: NCT00670423
Title: A Phase I Study Using Tacrolimus, Sirolimus and Bortezomib as Acute Graft Versus Host Disease Prophylaxis in Allogeneic Peripheral Blood Stem Cell (PBSC) Transplantation
Brief Title: A Study Using Tacrolimus, Sirolimus and Bortezomib as Acute Graft Versus Host Disease (GVHD) Prophylaxis in Allogeneic Peripheral Blood Stem Cell (PBSC) Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jennifer E. Schwartz (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jennifer E. Schwartz, Assistant Professor of Clinical Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0204; 0803-17 (Other: Indiana University IRB)
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Graft vs Host Disease; Peripheral Blood Stem Cell Transplantation; Transplantation, Homologous
Keywords: Tacrolimus; Sirolimus; Bortezomib; Acute Graft Versus Host Disease; Allogeneic Peripheral Blood Stem Cell Transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Tacrolimus; Sirolimus; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus as a continuous IV infusion will begin on day -3. (Levels will be monitored at least every 3 days to target 5-10 ng/mL)
  Other Names: Prograf®
Drug: Sirolimus — Sirolimus oral loading dose on day -3, followed by oral daily dose. (Levels will be monitored at least every 3 days to target 3-12 ng/mL)
  Other Names: Rapamune®
Drug: Bortezomib — Administered intravenously on day 0 (a minimum of 6 hours post-infusion of PBSC), and on day +3. The following dose levels will be used:
  Cohort 1 (3-6 pts): 1 mg/m2 on days 0 and +3
  Cohort 2 (3-6 pts): 1.3 mg/m2 on days 0 and +3
  Cohort 3 (3-10 pts): 1.6 mg/m2 on days 0 and +3
  Other Names: Velcade®

SUMMARY:
The purpose of this study is determine the highest dose of bortezomib, a new drug for graft-versus host disease prevention, that can be given in combination with sirolimus and Tacrolimus, without causing severe side effects. This research is being done because there is no treatment that is 100% effective in preventing graft versus host disease.

The goals of this study are to:

1. Collect peripheral blood stem cells (PBSCs) from donors for transplant.
2. Determine the largest possible dose of bortezomib that can be given to recipients with various blood cancers in a safe manner.
3. Monitor the recipient for risk of infection or side affects associated with the transplant.
4. Monitor the recipient for increased immunity following transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing myeloablative peripheral blood stem cell transplantation
* Have an HLA matched-related or matched-unrelated donor (9/10 antigen or allelic mismatch or 10/10 HLA match permitted).
* Hematological malignancy including patients with: AML, ALL, NHL, Hodgkin's Disease, CLL, CML, MDS and Multiple Myeloma
* Meeting institutional standard criteria for allogeneic PBSC transplantation

Exclusion Criteria:

* Patient has >Grade 2 peripheral neuropathy within 14 days before enrollment.
* History of autologous or allogeneic transplantation
* Evidence of HIV seropositivity
* Evidence of active infection
* Patients with cardiac dysfunction as described in the protocol
* Patients with hypersensitivity to bortezomib, boron or mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-05-16 (Actual); Primary Completion 2012-07-05 (Actual); Study Completion 2013-10-16 (Actual)

PRIMARY OUTCOMES:
To evaluate the maximum tolerated dose (MTD) of bortezomib in combination with tacrolimus and sirolimus as GVHD prophylaxis in patients undergoing myeloablative allogeneic peripheral blood stem cell transplantation. | Baseline through end of study

SECONDARY OUTCOMES:
To assess the toxicity of bortezomib | Baseline through end of study
To describe engraftment | Baseline through end of study
To describe the incidence of acute and chronic GVHD | Baseline through end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Schwartz, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States